CLINICAL TRIAL: NCT05169775
Title: A Single Centre, Prospective, Observational Study to Assess the Use of the Rehabilitation Tool, GripAble, in Patients With Upper Limb Spasticity Receiving Botulinum Toxin-A (BoNT-A) in the UK.
Brief Title: A Single Centre, Prospective, Observational Study to Assess the Use of the Rehabilitation Tool, GripAble, in Patients With Upper Limb Spasticity Receiving Botulinum Toxin-A (BoNT-A) in the United Kingdom (UK).
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52120-453
Record Dates: First submitted 2021-12-23; First posted 2021-12-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Upper Limb Spasticity (ULS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore how a rehabilitation tool (GripAble) could be used to monitor the effect of BoNT-A during an injection cycle and understand its potential value as a home rehabilitation tool in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiparesis with spasticity in the Primary Target Muscle Group (PTMG) for whom a decision to treat with BoNT-A has been made prior to inclusion in the study
* BoNT-A injection must be administered in the PTMG; injection into additional upper limb muscles must be based on investigator's judgment in line with the relevant Summary of Product Characteristics (SmPC)
* Naïve or non-naïve to BoNT-A treatment; if non-naïve, at least 4months elapsed after the last BoNT-A injection, of any marketed formulation prescribed in accordance to the relevant SmPC
* Must be able to use the GripAble tool and have access to the internet through wireless connection in the home setting
* Patients for whom the use of the GripAble tool aims to train:

  1. Wrist extension,
  2. Supination,
  3. Grip and release

Exclusion Criteria:

* Surgery on any upper limb or intrathecal baclofen therapy (ITB) for spasticity within the last 3 months
* Progressive neurological (e.g. Parkinson's Disease)
* Patients with no active muscle recruitment in the affected upper limb
* Patients with significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1 secondary care center in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Mean Physician Global Assessment (PGA) of treatment response scores in patients receiving BoNT-A for ULS during routine clinical practice. | At end of study (EOS) (between week 12 and week 20).
  The assessment of the treatment response to BoNT-A therapy will be recorded on a nine-point scale (range -4: markedly worse to +4: markedly improved).

SECONDARY OUTCOMES:
Changes from baseline in Modified Ashworth Scale (MAS) for Primary Target Muscle Group (PTMG). | At end of study (between week 12 and week 20).
Changes from baseline in MAS for Goal Attainment Scale (GAS)-T score | At end of study (between week 12 and week 20).
Changes from baseline in MAS for Passive Range of Motion (PROM) | At end of study (between week 12 and week 20)
Change from baseline in MAS for Active Range of Motion (AROM) | At end of study (between week 12 and week 20)
Changes from baseline in MAS | Time Frame: At end of study (between week 12 and week 20)
Changes from baseline in GAS-T score | At end of study (between week 12 and week 20
Changes from baseline in PROM | At end of study (between week 12 and week 20
Change from baseline in AROM | At end of study (between week 12 and week 20
Change from baseline in MAS by muscle group irrespectively of PTMG. | At end of study (between week 12 and week 20
Percentage of patients who achieved primary goal from GAS scaling | At end of study (EOS) (between week 12 and week 20)
Number of patients who set a primary goal per GAS | At baseline
Patient reported outcome of injection effectiveness on visual analogue scale (VAS) | Weekly basis up to end of study (between week 12 and week 20)
  A record of injection effectiveness on VAS (of 0 to 100 [bad to good]
Patients reported outcomes of treatment effects. | Weekly basis up to end of study (between week 12 and week 20
Dosing of BoNT-A administered | From baseline (first injection) to end of study (between week 12 and week 20)
  A record of dosing, BoNT-A brand, localisation method, dose per muscle will be recorded by the physician at each injection.
Target muscles injected | From baseline (first injection) to end of study (between week 12 and week 20)
  A record of the muscles injected at each injection.
Incidence of Adverse Events (AEs) or special situations | Up to 20 weeks
  Assessed according to incidence, seriousness, intensity, causality, outcome and action taken

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Hull University Teaching Hospital NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Abayomi Salawu, Sharah Abdul Mutalib, Anthony Cosgrove, Vadim Degtiar, Anne-Sophie Grandoulier, Helena MacCarthy-Ielo, Sharon Scott, Mario Ippolito. Single-Center, Prospective, Observational Study to Assess the Use the Rehabilitation Tool, GripAble, in Adults With Upper Limb Spasticity Receiving Botulinum Neurotoxin Type A in the UK. Toxicon, January 2024, Volume 237, Supplement 1, 107484.